CLINICAL TRIAL: NCT03592537
Title: Fentanyl Versus Midazolam as an Adjunct to Intrathecal Bupivacaine for Postoperative Analgesia in Children Undergoing Infraumbilical Surgery
Brief Title: Fentanyl Versus Midazolam as an Adjunct to Intrathecal Bupivacaine In Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa mahmoud Abd El Rady, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Fentanyl versus midazolam
Record Dates: First submitted 2018-03-28; First posted 2018-07-19 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Analgesia
Keywords: Fentanyl versus midazolam
MeSH Terms: interventions — Fentanyl; Midazolam; Bupivacaine

STUDY DESIGN:
Intervention Model Description: comparison of the effect of intrathecal fentanyl with the effect of intrathecal midazolam as postoperative analgesia in children undergoing infraumbilical surgery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care provider, Investigator, Outcomes Assessor) The trial will be planned that neither the doctors nor the patients will be aware of the group allocations. The study drugs will be prepared by an anesthesiologist not involved in performing the aneshesia, patient care or in data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fentanyl (Active Comparator): Group F: will receive intrathecal 0.5% bupivacaine (0.3 mg/kg) + (5ug) of fentanyl intrathecally
  Interventions: Drug: Fentanyl
- midazolam (Active Comparator): Group M: will receive intrathecal 0.5% bupivacaine (0.3 mg/kg) + 0.5 mg of midazolam intrathecally
  Interventions: Drug: Midazolam
- Bupivacaine (Placebo Comparator): Group B:intrathecal 0.5% bupivacaine (0.3 mg/kg)
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Fentanyl — The study drugs will be prepared by an anesthesiologist not involved in performing the anesthesia patient care or in data collection. Children will be randomly allocated into three groups of 30 children
  Other Names: sublimaze
  Arms: fentanyl
Drug: Midazolam — The study drugs will be prepared by an anesthesiologist not involved in performing the anesthesia, patient care, or in data collection. Children will be randomly allocated into three groups of 30 children
  Other Names: dormicum
  Arms: midazolam
Drug: Bupivacaine Hydrochloride — The study drugs will be prepared by an anesthesiologist not involved in performing the anesthesia, patient care, or in data collection. Children will be randomly allocated into three groups of 30 children
  Other Names: Bupivacaine
  Arms: Bupivacaine

SUMMARY:
The primary aim of the present study will be to compare the analgesic effect of addition of fentanyl or midazolam to intrathecal bupivacaine by using CHEOPS pain score (Children's Hospital Eastern Ontario Pain Scale) which is based on 6 criteria: crying, facial expression, child verbal expression, torso (body position), touching or grabbing at wound and legs position. Criterion 1 is given a score of 1-3, criteria 2 and 3 are given a score of 0-2 while criteria 4, 5 and 6 are given a score of 1-2; making the worst possible score 13 while the least possible score is 4. A total score ⩽ than 6 indicates adequate analgesia.

Secondary outcomes of study will be;

* is to compare the duration of postoperative analgesia.
* comparative assessment regarding time for first analgesic request ,total analgesic requirements.
* Hemodynamic changes or other adverse events will be recorded.

DETAILED DESCRIPTION:
Spinal anesthesia (SA) in pediatrics began to be used in the late nineteenth century in multiple procedures, with the priority for high-risk and former preterm infants, for its suggested protective role compared to the development of postoperative apnea with general anesthesia (GA) . Regional anesthesia offers several advantages over general anesthesia-blunts stress response to surgery, decreases intraoperative blood loss, lowers the incidence of postoperative thromboembolic events, and provides analgesia in early postoperative period .

Spinal anesthesia has been Proposed as a means to reduce postoperative complications especially apnea and postoperative respiratory dysfunction. Prolongation of pain relief can be accomplished by various adjuvants like opioids (morphine, fentanyl, ketamine and clonidine. However, each drug has its limitations and side effects, and the need for an alternative methods and drugs always exists. Of the several opioids available for neuro-axial administration, morphine and fentanyl remain the most commonly used agents. Because of the more lipophilic nature of fentanyl, it has a more rapid onset of action than morphine.

Intrathecal fentanyl produce profound analgesia by making direct contact with the substantia-gelatinosa of the cord and it also provides cephalad extend of sensorial block. The addition of intrathecal fentanyl to spinal anesthesia improves the intraoperative and the early postoperative quality of analgesia, relieves visceral pain and attenuates sympathetic activation during surgery . The addition of intrathecal midazolam gives the best prophylaxis against intraoperative and postoperative nausea and vomiting , also various studies have shown that the analgesic effect of intrathecal bupivacaine is enhanced by intrathecal midazolam without producing significant side effects.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-8years
* undergoing infra-umbilical surgery.

Exclusion Criteria:

* Children with a known history of bleeding diathesis,
* allergy to local anesthetics,

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | 24 hours
  CHEOPS pain score (Children's Hospital Eastern Ontario Pain Scale) which is based on 6 criteria: crying, facial expression, child verbal expression, torso (body position), touching or grabbing at wound and legs position. Criterion 1 is given a score of 1-3, criteria 2 and 3 are given a score of 0-2 while criteria 4, 5 and 6 are given a score of 1-2; making the worst possible score 13 while the least possible score is 4. A total score ⩽ than 6 indicates adequate analgesia.

SECONDARY OUTCOMES:
to compare the duration of postoperative analgesia. comparative assessment regarding time for first analgesic request ,total analgesic requirements and any adverse effects. | 24hour

CONTACTS AND LOCATIONS:
Overall Officials: Wesam N Ali, MD, Principal Investigator — lecturer
Locations (1):
- Pediatric hospital,assiut university, Asyut, Asyut Governorate, Egypt

REFERENCES:
- [Result] Chattopadhyay A, Maitra S, Sen S, Bhattacharjee S, Layek A, Pal S, Ghosh K. A study to compare the analgesic efficacy of intrathecal bupivacaine alone with intrathecal bupivacaine midazolam combination in patients undergoing elective infraumbilical surgery. Anesthesiol Res Pract. 2013;2013:567134. doi: 10.1155/2013/567134. Epub 2013 May 15. PMID 23762043
- [Result] Duman A, Apiliogullari S, Duman I. Effects of intrathecal fentanyl on quality of spinal anesthesia in children undergoing inguinal hernia repair. Paediatr Anaesth. 2010 Jun;20(6):530-6. doi: 10.1111/j.1460-9592.2010.03315.x. Epub 2010 Apr 23. PMID 20456062
- [Result] Dodawad R, G B S, Pandarpurkar S, Jajee P. Intrathecal Midazolam as an Adjuvant in Pregnancy-Induced Hypertensive Patients Undergoing an Elective Caesarean Section: A Clinical Comparative Study. Anesth Pain Med. 2016 Jul 26;6(5):e38550. doi: 10.5812/aapm.38550. eCollection 2016 Oct. PMID 27847698
- [Result] Lopez T, Sanchez FJ, Garzon JC, Muriel C. Spinal anesthesia in pediatric patients. Minerva Anestesiol. 2012 Jan;78(1):78-87. doi: 10.1111/j.1460-9592.2011.03769.x. Epub 2011 Dec 28. PMID 22211775
- [Result] Sanwatsarkar S, Kapur S, Saxena D, Yadav G, Khan NN. Comparative study of caudal clonidine and midazolam added to bupivacaine during infra-umbilical surgeries in children. J Anaesthesiol Clin Pharmacol. 2017 Apr-Jun;33(2):241-247. doi: 10.4103/0970-9185.209739. PMID 28781453